CLINICAL TRIAL: NCT01939171
Title: Conditioning of the Cadaver Donor by Thymoglobulin Administered to Reduce the Pro-inflammatory State After Brain Death.
Brief Title: Thymoglobulin in Cadaver Donor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Hospital de Santa Maria, Portugal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HULP- Nefro 001; 2009-013398-16 (EudraCT Number)
Record Dates: First submitted 2013-08-29; First posted 2013-09-11 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-09

CONDITIONS: Prevention of Kidney Injury Associated With Brain Death
Keywords: Thymoglobulin; Cadaver donor; Kidney injury brain death related
MeSH Terms: interventions — thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non treated (Placebo Comparator): Cadaver donor is cared and treated as usual protocol
- TREATED (Experimental): Cadaver donor receives one dose of thymoglobulin of 3 mg/kg iv in 2 hours after ganglia extraction and 3- 6 hours prior to organ procurement.
  Interventions: Drug: Thymoglobulin

INTERVENTIONS:
Drug: Thymoglobulin
  Arms: TREATED

SUMMARY:
To determine the efficacy and Security of Thymoglobuline in cadaveric donor Efficacy: To demonstrate that in cadaveric donor, Thymoglobuline diminished graft alloreactivity by decreasing expression of inflammatory markers in graft biopsies Security:To demonstrate that the administration of Thymoglobulin does not have side effects in renal recipients.

DETAILED DESCRIPTION:
This is randomized controlled Multicenter phase II clinical trial promoted by members from IdiPAZ. At least two hospital (La Paz and Santa Maria from Lisbon, will be involved. A per nature pilot study will recruit 10 cadaver donors from each hospital, and randomized half-to-half per center, for study and control groups.

The RCT initiated in 2009 and finished in 2013.

Cadaver donor from the study group will receive 3 mg/kg iv. Thymoglobulin 3-6 hours prior to organ procurement. The randomization process recruits 1:1 study/control donors.

Kidney biopsies will be taken from each kidney before transplantation to examine the expression of pro-inflammatory and HLA molecules (anti-DR, VCAM, ICAM, E-selectin) at tubular cells by immunohistochemical techniques under blinded conditions.

Recipients will be managed as usual and expressly followed up for one year, recording the incidence of delayed graft function and rejection and graft survival at the first year.

A comparison between the results obtained in kidney biopsies and patients transplanted in each group will permit differentiate whether Thymoglobulin administered in cadaver modifies the expression of antigens by kidney tubular cells and the results obtained with transplantation, in terms of graft function, rejection and survival.

ELIGIBILITY:
Inclusion Criteria:

* Accepted adults cadaveric donors for renal transplant from University Hospital La Paz( Madrid) and from University Hospital Santa Maria (Lisbon)
* Informed consent from relatives for including in the study

Exclusion Criteria:

* Known allergy to the rabbit proteins
* Non accepted grafts
* Family refusal to consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Efficacy of Thymoglobuline in cadaveric donor | 2 days
  To determine the efficacy of Thymoglobuline in cadaveric donor Efficacy: To demonstrate that in cadaveric donor, Thymoglobuline diminished graft alloreactivity by decreasing expression of inflammatory markers(determining HLA-DR,VCAM-1, ICAM-1 expressions by immunohistochemistry in graft biopsies), and the rates of delayed graft function and cellular/humoral rejection demonstrated by biopsy.
Security of Thymoglobuline in cadaveric donor | 1 day
  Estimated by general and particularly hemodynamic tolerance to thymoglobulin infusion.

SECONDARY OUTCOMES:
Incidence of acute rejection in the recipients | 3 moths
  To demonstrate that in cadaveric donors, Thymoglobuline tends to decrease the incidence of acute rejection demonstrated by kidney biopsy.
Incidence of delayed graft function in the recipients. | 1 month
  To demonstrate that in cadaveric donors, Thymoglobuline tends to decrease the incidence of DGF estimated by the necessity of dialysis after transplantation.
Composite of incidence of graft function and general effects in the recipients. | 1 year
  To demonstrate that Thymoglobuline administered in cadaveric donors does not have neither repercussion on graft function nor side effects in renal and liver recipients.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Jimenez, MD, PhD, Principal Investigator — Hospital Universitario La Paz; Maria Lopez-Oliva, MD, Principal Investigator — Hospital Universitario La Paz; Rui Mayo, MD, Principal Investigator — Hospital Santa Maria, Portugal
Locations (2):
- Hospital Santa Maria, Lisbon, Lisbon District, Portugal
- Hospital Universitario La Paz, Madrid, Madrid, Spain

REFERENCES:
- See also: Medical Research Institute — http://www.idipaz.es/